CLINICAL TRIAL: NCT01680250
Title: An Open-label, Prospective Clinical Trial to Evaluate the Effectiveness and Safety of Sirolimus to Reduce Cyst Growth in ADPKD Patients With Massive Polycystic Liver
Brief Title: Sirolimus for Massive Polycystic Liver
Acronym: SILVER
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SILVER
Record Dates: First submitted 2012-08-30; First posted 2012-09-07 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Polycystic Kidney Diseases
Keywords: Total liver volume; Liver cyst
MeSH Terms: conditions — Polycystic Kidney Diseases | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sirolimus (Experimental): Sirolimus administration group starting dose: 2mg/day target trough level: 4-10 ng/dL
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Sirolimus administration for 12 months followed by conventional therapy alone for additional 12 months
  Other Names: Rapamune

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of Sirolimus in reducing liver volume in autosomal dominant polycystic kidney disease.

DETAILED DESCRIPTION:
Autosomal dominant polycystic kidney disease (ADPKD) is one of the most common causes of end stage renal disease (ESRD), affecting an estimated 0.2% of population. Of ADPKD patients, 58% in 15-24 year, 85% in 25-34 year, and 94% in 35-46 year olds suffer from polycystic liver in addition to polycystic kidneys. Several anti-proliferative drugs have been used in clinical trials to stop cyst growth both in liver and kidneys. Among them, octreotide and sirolimus have been shown to be one of the most promising drugs to reduce cyst volume. Sirolimus already has been used as one of the most potential oral immunosuppressants. Moreover, the serum trough level is quite easy to measure. Sirolimus is the mTOR inhibitor that has been proven to be effective in reducing cyst growth both in animal models. However, its efficacy and safety is not well proven in previous studies. This is a open-label, prospective study to evaluate the effectiveness and safety of Sirolimus to reduce cyst growth in ADPKD patients with massive polycystic liver.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65
* Patients diagnosed as ADPKD based upon the unified criteria for ultrasonographic diagnosis of ADPKD
* Polycystic liver with total liver volume > 2500 mL or symptomatic polycystic liver
* Estimated glomerular filtration rate (IDMS-traceable MDRD equation) >= 30 mL/min/1.73m2

Exclusion Criteria:

* Concomitant systemic renal parenchymal or urinary tract disease (random urine albumin-to-creatinine ratio > 500 mg/g)
* WBC < 4,000/uL, platelet < 100,000/uL, or hemoglobin < 10.0 g/dL
* Diabetes mellitus, cancer, or psychiatric disorder
* Increased liver enzymes (2-fold above normal value)
* Hypercholesterolemia (fasting cholesterol > 200mg/dL) or hypertriglyceridemia (>150 mg/dL) not controlled by lipid lowering therapy
* Infection with hepatitis B, C, HIV
* Any condition that could prevent full comprehension of the purpose and risks of the study
* Pregnant or lactating women or fertile women without effective contraception
* History of intervention, such as cyst aspiration or embolization in past 1 year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-09 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Total liver volume | 12 months
  Change in total liver volume

SECONDARY OUTCOMES:
Total liver volume | 24 months
  Change in total liver volume
Total kidney volume | 12 month
  Change in total kidney volume
Estimated glomerular filtration rate | 12 month
  Change in estimated glomerular filtration rate
Urinary biomarker | 12 month
  Urinary biomarker level
Total kidney volume | 24 month
  Change in total kidney volume
Estimated glomerular filtration rate | 24 month
  Change in estimated glomerular filtration rate
Urinary biomarker | 24 month
  Urinary biomarker level

OTHER OUTCOMES:
Abdominal pain | 12month
  Abdominal pain quantified by Visual Analog Scale
Abdominal pain | 24 month
  Abdominal pain quantified by Visual Analog Scale
Infection | 24 month
  Incidence of infection event during study time
Hospitalization | 24 month
  Incidence of hospitalization due to adverse events during study time
Drop out | 24 month
  Incidence of discontinuation of study drug due to serious adverse events during study time

CONTACTS AND LOCATIONS:
Overall Officials: Curie Ahn, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea